CLINICAL TRIAL: NCT06451692
Title: Prioritising Patient Medication Review: Hospitals Reaching Out (PriPMed)
Brief Title: Prioritising Patient Medication Review: Hospitals Reaching Out
Acronym: PriPMed
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SHS-Pharm2 - 2024
Record Dates: First submitted 2024-05-28; First posted 2024-06-11 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Medication Review; Polypharmacy; General Practitioners; Interdisciplinary Communication; Clinical Pharmacy
Keywords: Multi-morbidity; Medication review; Dementia; Clinical Fragility scale; Hospital to home transition; Polypharmacy
MeSH Terms: conditions — Dementia | interventions — Pharmacists

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The clinical pharmacist will assess the patient's medication, and perform interviews with the patient and/or the patient's attorney-in-fact. Potential medical recommendations will be discussed with the treating hospital clinician and the clinical pharmacist, and a medication plan will be developed together with the patient or the patient's attorney-in-fact. The GPs will be informed through optimized discharge summaries.
  Interventions: Other: Clinical pharmacist
- Control group (No Intervention): Patients in the control group receive standard care without a clinical pharmacist involved in the healthcare team at ward level. Standard care consists of usual treatment from a team of hospital physicians, nurses, nurse assistants, and as needed occupational therapists, physiotherapist, and clinical dieticians. Hospital physicians and/or nurses might perform patient counselling about medication treatment during hospitalization

INTERVENTIONS:
Other: Clinical pharmacist — The clinical pharmacist calls the patients' GP 90 days after discharge for follow-up
  Arms: Intervention group

SUMMARY:
To examine the effect of a cross-sectoral medication review intervention to admitted multi-morbid, polypharmacy patients aged 65+ at SHS in two settings; an acute admission unit (typical admission time < 48 hours) and a medical outpatient setting (patients routinely visits for follow-up, diagnosis or treatment, but do require a bed or overnight care).

DETAILED DESCRIPTION:
Lack of medication treatment coordination among especially multi-morbid patient's results in suboptimal medication treatment, adverse effects, increased use of resources, hospital admissions and premature death. Further, an aging population is a challenge to healthcare systems worldwide as older adults are vulnerable to non-communicable diseases and multi-morbidity. The age distribution varies across Denmark creating demographic inequality with a higher proportion of elderly in several municipalities in Southern Jutland and on a national level, the population aged 70+ already accounts for more than a third of all hospital days.

As the population ages, the concept of frailty becomes increasing in the provision of health care to an ageing population, and the Clinical Frailty Scale (CFS) can be used as a judgement-based frailty tool to evaluate specific domains including comorbidity, function, and cognition to generate a frailty score. In addition, an attempt to detect patients at high risk of medication errors is the Medicine Risk Score (MERIS) where acutely admitted patients are allocated into low and high risk of potential ADEs by predefined detection limits. Further, These components will be used to determine

In addition, an understudied patient group within polypharmacy and PIPs, are patients with dementia creating inequality among patient groups. The use of polypharmacy and Potential Inappropriate Prescribing are widespread in this patient group, and dementia is well-known to have a negative effect on overall mortality, which demonstrates the need for interventions to improve medication treatment in people with dementia. Intervention studies have examined the effects of pharmacist-led medication reviews in different hospital settings with various outcomes, but no exact model for prioritising patient medication review exists. Thus, there is a need to identify patients who will benefit most from a medication review in terms of outcomes, such as readmission, emergency department and general practitioner contacts. The aim of this project is to examine the effect of a cross-sectoral medication review between a clinical pharmacist and a medical specialist in coordination with the General Practitioner (GP), including patients from Hospital Sønderjylland, University Hospital of Southern Denmark (SHS).

ELIGIBILITY:
Inclusion Criteria:

* all hospitalized patients who are prescribed at least seven medications specified in the Electronic Patient Journal (EPJ) at admission

Exclusion Criteria:

* terminal patients or patients with a short life expectancy, patients residing in another region, patients who are discharged on the day of inclusion, and finally patients who do not speak Danish.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Readmission and emergency department rate. | Up to thirty days after discharge
  The number of acute readmissions and emergency department visits between 4 hours and 30 days after discharge from the index hospital stay in the intervention group compared with the control group. As a "yes" or "no" and a time-to-event. Potential readmissions are assessed through the electronic patient journal.

SECONDARY OUTCOMES:
Acute admission | Up to 90 days after discharge
  Time to first acute admission after discharge from index hospital stay for the intervention and control group (up to 90 days follow-up). As a "yes" or "no" and a time-to-event. Potential acute admissions are assessed through the electronic patient journal.
Mortality | 30 and 90 days after discharge
  The mortality rate after 30 and 90 days respectively after discharge will be evaluated. As a "yes" or "no" and a time-to-event. The mortality will be identified from patient journals.
GP contacts | Up to 90 days after discharge
  The GP visit rate (number) will be identified at a follow-up telephone contact with the GP 90 days after discharge. As a "yes" or "no" to GP contact within the time frame and a time-to-event related to "yes".
Implementation rate | Up to 90 days after discharge
  The implementation rate (number) of pharmacist recommendations and potential medication changes from the medication review made by the GP will be identified, 30 and 90 days respectively after index hospital stay. Each recommendation will be evaluated as a "yes", "no", "partly" or "unsure", where "partly" or "unsure" requires additional free text information to support the evaluation. The information will be obtained from the patients' shared medication record
Compliance with medical treatment | Up to 90 days after discharge
  Patient compliance with their medical treatment will be obtained from the patients' shared medication record with information on all patient purchases of prescribed medications. As a "yes", "no", "partly" or "unsure".

OTHER OUTCOMES:
Patient satisfaction with the intervention | 7 to 10 days after discharge
  Patients' satisfaction and experience with the medication review and intervention are explored through a smaller sample of intervention patients (approx. 25%, 50 patients) using an evaluation survey and a 5-likert scale. The evaluation will be conducting through telephone by the project manager, who will follow a structured evaluation survey and register the patients reply continuously in an online survey form in RedCap.
Evaluation of the collaboration among clinical pharmacists, medical specialists, and GPs | 10 months after the randomization of the first participant in each setting an online survey link will be sent clinical pharmacists, medical specialists, and GPs
  The evaluation of the collaboration will be explored through a survey to clinical pharmacists, medical specialists, and GPs. The main focus are the collaboration with the GP and medical doctors; potential barriers to a fruitful collaboration in the team of clinical pharmacist, medical specialist and the GP; the feasibility of the intervention with pharmacist-led medication review to admitted patients, and the experience with the optimized discharge summary containing pharmacist interventions from medication reviews. A 5-likert scale will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Sygehus Sønderjylland, Aabenraa, Southern Denmark, Denmark